CLINICAL TRIAL: NCT02871648
Title: The Role of Minerelocorticoid Receptor on Modulating Aldosterone Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gordon H. Williams, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2015P001664
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy
MeSH Terms: interventions — Fludrocortisone; fludrocortisone acetate; Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo prepared by Investigational Drug Services at Brigham and Women's Hospital
  Interventions: Drug: Placebo
- Fludrocortisone (Active Comparator): Subjects will receive 0.1 mg of fludrocortisone (Florinef) on one of three study days.
  Interventions: Drug: Fludrocortisone
- Epleronone (Active Comparator): Subjects will receive 100 mg of epleronone on one of three study days.
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Placebo — Placebo prepared by Investigation Drug Services at Brigham and Women's Hospital
  Arms: Placebo
Drug: Fludrocortisone — Fludrocortisone 0.1 mg
  Other Names: Florinef
  Arms: Fludrocortisone
Drug: Eplerenone — Epleronone 100 mg
  Other Names: Inspra
  Arms: Epleronone

SUMMARY:
The purpose of this research protocol is to determine if the same effects are observed in vivo in humans using a similar approach. Demonstrating that mineralocorticoid acts on zona glomerulosa cells to regulate aldosterone production in a short feedback loop would provide important insight into hormone regulation, and explain variability in pathophysiologic states such as hypertension and cardiovascular diseases.

DETAILED DESCRIPTION:
In order to provide additional evidence indicating the presence of functional and in order to provide additional evidence indicating the presence of functional mineralocorticoid receptors (MR) on zona glomerulosa (ZG) cells, the investigators propose the following protocol in healthy volunteers. The investigators will evaluate aldosterone and cortisol production in response to an angiotensin II infusion after three separate test conditions: 1) placebo, 2) following a single dose of fludrocortisone, and 3) following a single dose of eplerenone (a MR antagonist).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy, with no prior history of hypertension, no family history of hypertension, diabetes, stroke or cardiac disease in first-degree relatives before the age of 70 years and have an average (two measurements) blood pressure of <130/89 mm Hg and >100/50 mmHg at the screening visit.
* All subjects will have body mass index 19-25 kg/m2.
* Subjects must have normal laboratory values for: Complete blood count; serum creatinine, sodium, potassium, glucose, liver enzymes; urinalysis; negative urine HCG in women; normal ECG

Exclusion Criteria:

* Alcohol intake >12oz per week, as well as tobacco or recreational drug use.
* Any subject with a history of coronary disease, diabetes, hypertension, stroke, kidney disease, or illness requiring overnight hospitalization in the past 6 months will be excluded from the study.
* Subjects taking any prescription medications (with the exception of birth control pills) or herbal medications will be excluded.
* Because of the unknown risk of infused angiotensin II in pregnancy, women who are pregnant will be excluded from study and all women will be screened for pregnancy by quantitative serum hCG measurement on the day of each CCI admission.
* Women currently breastfeeding will also be excluded from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01; Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Serum aldosterone after angiotensin II infusion | 5 days
  Aldosterone levels after 30 mins AngII infusion

SECONDARY OUTCOMES:
Serum aldosterone after cosyntropin infusion | 5 days
  Aldosterone levels after 30 mins cosyntropin infusion
Serum cortisol after angiotensin II infusion | 5 days
  Cortisol levels after 30 mins AngII infusion
Serum cortisol after cosyntropin infusion | 5 days
  Cortisol levels after 30 mins cosyntropin infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Williams, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braley LM, Williams GH. Rat adrenal cell sensitivity to angiotensin II, alpha-1-24-ACTH, and potassium: a comparative study. Am J Physiol. 1977 Nov;233(5):E402-6. doi: 10.1152/ajpendo.1977.233.5.E402. PMID 200147